CLINICAL TRIAL: NCT02715089
Title: Single Center, Single Arm, Open Study, to Explore and Evaluate the Precise Treatment in Hepatobiliary Cancers(PTHBC)
Brief Title: Precise Treatment in Hepatobiliary Cancers (PTHBC)
Acronym: PTHBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: 3D Medicines (Industry)
Responsible Party: Sponsor
Other Study IDs: PM1503
Record Dates: First submitted 2016-02-28; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Liver Neoplasms; Biliary Tract Neoplasms; Hepatobiliary Neoplasms
Keywords: NGS; Liver Neoplasms; Biliary Tract Neoplasms; Hepatobiliary Neoplasms
MeSH Terms: conditions — Liver Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The samples, both tissue(s) and blood of patients should be provided for the next-generation sequencing (NGS) test before screening.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Precise treatment: All patients should accept next-generation sequencing (NGS) test before treatment.
  Interventions: Genetic: Precise treatment

INTERVENTIONS:
Genetic: Precise treatment — During screening stage, all patients should accept next-generation sequencing (NGS) test.

SUMMARY:
The purpose of this study is to explore the precise treatment in hepatobiliary cancer patients and evaluate drug safety, progression free and overall survival. This trial study is based on genetic tests, then therapeutic target drugs are administered according to the genetic test reports. Patients with genetic abnormalities (such as mutations, amplifications, or translocations) may benefit from precise treatment which targets particular genetic abnormality. The identifications of these genetic abnormalities may help treat hepatobiliary cancer patients better.

DETAILED DESCRIPTION:
The genetic tests are performed for the eligible subjects in this study, then therapeutic target drugs are administered according to the genetic test reports. While the precise treatments, follow-ups are conducted to evaluate the efficacy and safety of the target drugs for the subjects, until the overall survival.

Study Type: Non-Interventional. Masking: Open Label.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65, male or female.
* Radiologically and pathologically confirmed as hepatobiliary cancers with stage IV.
* Palliative care as the preferred.
* The result of next-generation sequencing (NGS) test show the patient has gene mutation and also can be treated by the right commercial products that have been approved by the China Food and Drug Administration (CFDA) or the Food and Drug Administration (FDA).
* ECOG performance status 0-2.
* Life expectancy ≥3 months.
* Voluntarily participate in the study and agree to sign informed consent form.

Exclusion Criteria:

* Hepatobiliary cancer patient with stageI-III, or with any of the following items will not be eligible for screening.Such as, suitable for the treatment of radical resection, radical resection but evaluation unmeasurable.
* The result of NGS test show the patient has no gene mutation, or has gene mutation but no medicine.
* ECOG performance status ≥ 3.
* Female patients who are pregnant or not using a contraceptive method of birth control.
* History or presence of serious cardiovascular or cerebrovascular abnormalities.
* Abnormalities of the hepatic or renal functions, such as jaundice, ascites, bilirubin ≥ 1.5×ULN, alkaline phosphatase ≥ 3×ULN, persistent protein urine≥ grade 3 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0), creatinine ratio > 3.5g/24 hours, renal failure.
* Persistent infection > grade 2 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0).
* Patient has underwent a major operation 4 weeks prior to screening or has not yet recovered from the operation.
* Patient with epilepsy, known or untreated brain metastases.
* The presence of wounds, ulcers or fractures that can not be healed, or with a past history of transplantation.
* The presence of bleeding events ≥grade 3 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0) , present evidence or past history of coagulation dysfunction disorders.
* Known human immunodeficiency virus (HIV) infection history.
* Patient with drug abuse or unstable compliance.
* The presence of unresolved toxicity caused by any previous treatment/operation > grade 1 (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTC-AE] v4.0), except alopecia, anemia or hypothyroidism).
* Investigator consider that the patient should not be enrolled in this study by careful assessment.
* The subjects participate in any other clinical trial in the meantime.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects : Hepatobiliary Cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | 6 weeks
  Defined as the percentage of patients whose tumors have a complete or partial response to treatment (RECIST v1.1) .
Progression-free survival (PFS) | 8 months
  Progression-free survival (PFS) is the time that passes from the day in which the patient is enrolled in the trial until the date on which disease "progresses" or the date of death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Through study completion, an average of 1 year.
  Overall survival (OS) is the duration from the day in which the patient is enrolled in the trial until the date of death from any cause.
Duration of Response (DOR) | 6 months
  Duration of Response (DOR) is the duration from the first assessment of the tumor was CR or PR to the time that the first assessment for PD (Progressive Disease) or date of death from any cause.
Disease control rate (DCR) | 6 weeks
  Defined as the percentage of patients whose tumors have a complete or partial response，or stable disease to treatment (RECIST v1.1).
Adverse Drug Reaction (ADR)/Adverse Event (AE) | Through study completion, an average of 2 years.
  Patients with treatment-related adverse events as assessed by CTC-AE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Tao Zhao, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The data have the gene mutations information of patients.

REFERENCES:
- [Derived] Lin J, Shi J, Guo H, Yang X, Jiang Y, Long J, Bai Y, Wang D, Yang X, Wan X, Zhang L, Pan J, Hu K, Guan M, Huo L, Sang X, Wang K, Zhao H. Alterations in DNA Damage Repair Genes in Primary Liver Cancer. Clin Cancer Res. 2019 Aug 1;25(15):4701-4711. doi: 10.1158/1078-0432.CCR-19-0127. Epub 2019 May 8. PMID 31068370